CLINICAL TRIAL: NCT03291899
Title: Phase II Trial of Infusional 5 FLUOROURACIL, LEUCOVORIN, OXALIPLATIN AND IRINOTECAN (FOLFIRINOX) in First Line Treatment of Advanced Biliary Tract Cancers
Brief Title: Trial of Infusional FOLFIRINOX in First Line Treatment of Advanced Biliary Tract Cancers
Acronym: FBI-TRAC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Shouki Bazarbashi, section Head,Medical oncology, King Faisal Specialist Hospital & Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC 2161 099
Record Dates: First submitted 2017-09-21; First posted 2017-09-25 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — folfirinox

STUDY DESIGN:
Intervention Model Description: Simon 2-stage optimum design Model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental single arm (Experimental): Chemotherapy using the FOLFIRINOX regimen will be given every 2 weeks for a total of 12 cycles. FOLFIRINOX consist of:
  1. Oxaliplatin-85 mg/m2 IV Day 1
  2. Leucovorin-400 mg/m2 IV Day 1
  3. Irinotecan-180 mg/m2 IV Day 1
  4. Fluorouracil (FU)-400 mg/m2 IV bolus Day 1
  5. Fluorouracil 2400 mg/m2 infused over 46 hours starting day 1
  Interventions: Combination Product: FOLFIRINOX

INTERVENTIONS:
Combination Product: FOLFIRINOX — combination chemotherapy using Oxaliplatin, Irinotecan, Leucovorin and Fluorouracil, given every 15 days for a total of 12 cycles

SUMMARY:
This study is to evaluate the response rate and toxicity profile of infusional 5 fluorouracil, leucovorin, oxaliplatin and irinotecan (FOLFIRINOX) in first-line treatment of advanced biliary tract cancers and also to assess progression free survival and overall survival of FOLFIRINOX in first line treatment of advanced biliary tract cancers

DETAILED DESCRIPTION:
Biliary tract carcinomas (BTCs) are invasive adenocarcinomas that arise from the epithelial cells of the biliary tree, which comprises intrahepatic and extrahepatic bile ducts, and the gallbladder. Even though BTCs are considered as rare tumors, they represent about 30% of the total primary liver cancers with an incidence rate close to that of hepatocellular carcinoma. Approximately 1200 new cases in the United Kingdom and 9000 in the United States are diagnosed annually. The Saudi Cancer Registry reported 911 case of gall bladder cancer, 318 intrahepatic cholangiocarcinoma and 574 extrahepatic cholangiocarcinoma between 1994 and 2009. Unfortunately, only a minority of patients diagnosed with these aggressive tumors present at an early resectable stage, and disease recurrence rates are high despite curative-intent surgery

The prognosis of patients with advanced biliary tract cancers is poor and median survival for those undergoing supportive care alone is short. Systemic chemotherapy is increasingly being applied in cases of advanced biliary tract cancers. A benefit for chemotherapy over best supportive care alone was suggested in a trial that randomly assigned 90 patients with advanced pancreatic or biliary cancer (37 with bile duct cancer) to fluorouracil (FU)-based systemic chemotherapy or best supportive care alone with median survival of 6 months for chemotherapy versus 2.5 months for best supportive care.

Different drugs has demonstrated activity in BTCs, including fluoropyrimidines, gemcitabine, cisplatin, and oxaliplatin. A pooled analysis from Eckel et al. that evaluated 104 trials with 2810 patients, has established gemcitabine combined with platinum compounds as the provisional standard of chemotherapy in advanced biliary tract cancer.

In a randomized phase two study of 51 patients, Kornek et al, established the efficacy of mitomycin in combination with gemcitabine or capecitabine in previously untreated patients with advanced biliary tract cancers. Mitomycin and capecitabine was associated with superior complete response rate (31% vs 20%), median progression free survival (5.3 months vs 4.2 months), and overall survival (9.25 months and 6.7 months). The EORTC 40955 trial randomized patients with BTCs to high dose 5FU vs combination of 5-FU, Leucovorin and cisplatin. The results showed that cisplatin and fluorouracil was more active than high-dose fluorouracil in terms of overall response rates (19% and 7.1%, respectively) and overall survival (8 months and 5 months, respectively), but progression free surviva; was similar in both treatment arms (3.3 months).

The randomized, controlled, phase three ABC-02 study, which enrolled 410 patients with locally advanced or metastatic cholangiocarcinoma, gallbladder cancer or ampullary cancer, demonstrated that the combination of gemcitabine and cisplatin improved overall and progression free survival by 30% over gemcitabine alone. Median overall survival was 11.7 months vs 8.1 months (HR, 0.64; 95% confidence interval, 0.52-0.80; p˂.001), and progression free survival was 8 months (HR, 0.51; 95% confidence interval, 0.51-0.77; p˂.001), both in favor of the combination arm. Although the rate of neutropenia was higher in the group receiving gemcitabine and cisplatin, there was no significant difference in the rate of neutropenia-associated infections between the 2 arms. Okusaka et al also reported similar findings in a phase two randomized study of 84 patients with advanced biliary tract cancers. Based on these results, the combination of gemcitabine and cisplatin is considered to be the standard of care for first-line chemotherapy for patients with advanced or metastatic biliary tract cancers.

Triple-drug chemotherapy regimens also have been shown to be effective in patients with advanced biliary tract cancers, albeit in a very small number of patients. The phase three trial that evaluated fluorouracil, leucovorin and etoposide versus fluorouracil cisplatin and epirubicin didn't show one regimen to be significantly superior with respect to overall survival (12 months vs. 9 months, respectively) in patients with advanced biliary tract cancers, although the trial was underpowered to detect such a difference.

In a phase two trial, the combination panitumumab, a monoclonal anti-epidermal growth factor receptor antibody, with gemcitabine and irinotecan showed encouraging efficacy with good tolerability in patients with advanced cholangiocarcinoma, with 5-month progression free survival rate of 69%.The median progression free survival and overall survival were 9.7 months and 12.9 months, respectively.

Results from the randomized phase three PRODIGE trial evaluating the combination of 5-Fluorouracil, Leucovorin, oxaliplatin and Irinotecan (FOLFIRINOX) versus gemcitabine alone in patients with metastatic pancreatic cancer and good performance status showed dramatic improvements in both median PFS (6.4 vs 3.3 months; P˂ .001) and median OS (11.1 months vs. 6.8 months; P˂ .001). Because of these strong results the National comprehensive cancer network (NCCN) and many other societies added FOLFIRINOX as a preferred, category 1 recommendation for first line treatment of good performance status patients with metastatic pancreatic cancer in 2011.

There are, however, some concerns about the toxicity of FOLFIRINOX regimen. In the PRODIGE trial, some of the grade 3 and 4 toxicity rates that were significantly greater in the FOLFIRINOX group than in the gemcitabine group were 45.7% for neutropenia, 12.7% for diarrhea, and 9.1 % for thrombocytopenia and 9% for sensory neuropathy.

Despite the high levels of toxicity, no toxic deaths have been reported. Furthermore, the PRODIGE trial determined that, despite this toxicity, fewer patients in the FOLFIRINOX group than in the gemcitabine group experienced a degradation in their quality of life at 6 months (31% vs. 66%,p ˂ .001). A more detailed analysis of the quality of life of patients in this trial has been published and shows that FOLFIRINOX maintained and even improved quality of life more than gemcitabine did.

Based on the above data, the investigators designed this phase two study of the efficacy and toxicity of FOFIRINOX regimen in first line treatment for patients with advanced biliary tract cancers. If the investigators achieved encouraging results, this regimen should then be compared with the standard combination of gemcitabine and cisplatin in future phase three trials.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed locally advanced (irresectable) or metastatic biliary tract cancers.
2. Measurable disease. Defined as tumor that have uni or bi dimensional measurement not less than 1.5 cm on any dimension.
3. Age ≥ 18 years.
4. Signed written informed consent before enrolment.
5. No prior chemotherapy or anti-neoplastic therapy other than radiotherapy more than 4 weeks prior to enrolment and to areas other than the measurable disease.
6. Patients of either sex or child bearing age must be willing to use adequate contraceptive measures during the study and for 6 months after treatment.
7. Life expectancy of 6 months or more.
8. Eastern Cooperative Oncology Group performance status of 0-1.
9. Adequate renal function: creatinine within normal institutional range.
10. Adequate hepatic function: Total bilirubin within normal institutional limits, serum aspartate aminotransferase and alanine aminotransferase levels ≤2.5 times the institutional upper limit of normal or ≤ 5 times the institutional upper limit of normal of elevated because of liver involvement.
11. Adequate hematological values: leukocyte count ≥3.0 x 109/L, an absolute neutrophil count ≥1.5 x 109/L, a platelet count ≥100 x 109/L.

Exclusion Criteria:

1. Known or suspected dihydropyrimidine deficiency.
2. Presence of central nervous system metastasis.
3. Previous malignancy within 5 years, except adequately treated non melanomatous skin cancer or in situ cervical cancer.
4. Severe cardiovascular disease (congestive heart failure New York Heart Association class three or four, unstable angina pectoris, myocardial infarction or significant arrhythmias).
5. Psychiatric or mental disorder, precluding understanding of the information of the trial related topics and giving valid informed consent.
6. Active uncontrolled infection.
7. Pregnant patients (confirmed by β-Human chorionic gonadotrophin test where appropriate).
8. Serious underlying medical condition (in the judgement of the investigator) which could impair the ability of the patient to participate in the trial.
9. Any psychological, familial, geographic or social circumstances which could impair the patient's ability to participate in the trial and comply with follow up.
10. Treatment with other experimental drugs within 30 days of entry into the trial.
11. Treatment with other anti-cancer therapy.
12. Known hypersensitivity to any of the study drugs.
13. Breast feeding
14. Legal incapacity.
15. Patients with a known diagnosis of HIV infection.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Response rate | 3 year
  Evaluate the response rate using RECIST 1.1 criteria

SECONDARY OUTCOMES:
progression free survival | 4 years
  calculated from day 1 of chemotherapy till either progression, death or date of last follow up whichever comes first
overall survival | 4 years
  calculated from day 1 of chemotherapy till either death or date of last follow up whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Shouki Bazarbashi, Principal Investigator — King Faisal Specialist Hospital and Research cente
Locations (1):
- king Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Result] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404